CLINICAL TRIAL: NCT01593007
Title: REGIONAL LUNG VENTILATION DISTRIBUTION AMONG INDIVIDUALS WITH CHRONIC HEART FAILURE AFTER AN INSPIRATORY MUSCLE TRAINING PROGRAMM: A RANDOMIZED CONTROLLED CLINICAL TRIAL
Brief Title: Inspiratory Muscular Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Ciência e Tecnologia de Pernambuco (Other)
Responsible Party: Principal Investigator, Daniella Cunha Brandao, PhD, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tese02
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2011-10

CONDITIONS: Heart Failure
Keywords: Heart failure; respiratory muscles; optoelectronic plethysmography
MeSH Terms: conditions — Heart Failure | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inspiratory Muscle Training (Experimental): Inspiratory Muscle Training
  Interventions: Other: Inspiratory muscle training
- Control group (Placebo Comparator): Patients from the control group were also assessed weekly to ensure homogenization of the learning effect for the manometer maneuver.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Inspiratory muscle training — All participants were instructed to use a Threshold® trainer for 30min a day, seven times a week over 12 consecutive weeks.10 Patients in the Control Group used a Threshold ® device without resistance, making them blind to the treatment. For the treatment group, inspiratory resistance of the Threshold® trainer was 30% of MIP, adjusted on a weekly basis to remain constant.
  Arms: Inspiratory Muscle Training
Other: Control group — Patients from the control group were also assessed weekly to ensure homogenization of the learning effect for the manometer maneuver.
  Arms: Control group

SUMMARY:
Objectives: To evaluate regional lung ventilation distribution in patients suffering from chronic heart failure (CHF) after completing inspiratory muscle training (IMT) and correlate it with functional capacity and quality of life among these individuals. Methods and Results: Nineteen CHF patients were randomly assigned to two groups: Control and IMT. Before and after muscle training, subjects were submitted to assessment protocol for respiratory muscles, digital spirometry, optoelectronic plethysmography (OEP), the six-minute walk test (6MWT) and a quality of life questionnaire (MLHFQ). There was no difference in lung function following the 12-week training period in either group. However, the IMT group showed an increase in actual and predicted MIP, higher MLFHQ score and greater distance walked in the 6MWT, as well as a reduction in the Borg scale after the 6 MWT in relation to the control. For the OEP, IMT group members exhibited higher values for total chest wall volume (Vcw), abdominal rib cage volume (Vrc,a) and abdominal volume (Vab) when compared to the control. Conclusions: For patients with CHF, IMT proved efficient in improving muscle strength, functional capacity and quality of life. The present study also analyzed the distribution behavior of lung volumes for the thoracoabdominal system in this population, showing that larger abdominal rib cage and abdomen volumes may result in more effective diaphragmatic contraction.

ELIGIBILITY:
Inclusion Criteria:

* sedentary adults diagnosed with functional class II and II CHF in accordance with the New York Heart Association (NYHA);
* in stage B or C according to American College of Sports Medicine guidelines;
* with left ventricle ejection fraction lower than 45% (evaluated by echocardiogram in a period ≤ 1 year);
* cardiomegaly confirmed by increased left ventricle end-diastolic (LVDD) and end-systolic diameter (LVESD) associated with a cardiac index (CI) >0.5 according to chest X-rays;
* inspiratory muscle weakness (MIP <70% of predicted values);
* clinical stability with no change in medication for at least three months and sedentary (no regular physical activity performed in the previous six months or not accumulating 30 minutes or more of moderate physical activity - 3 to 6 METs - on most week days).

Exclusion Criteria:

* patients exhibiting unstable angina, myocardial infarction or prior heart surgery up to three months before beginning the investigation;
* orthopedic, infectious or chronic metabolic diseases;
* treatment with steroids, hormones or chemotherapy;
* ratio between forced expiratory volume in one second and forced vital capacity (FEV1/FVC) < 70% of predicted, characterizing an obstructive respiratory disorder;
* respiratory diseases, smokers and ex-smokers with a history of cigarettes/day for more than 10 years.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-06; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Respiratory muscles | 3 months
  In order to evaluate inspiratory muscle strength, a digital manometer was used (MVD-300, Globalmed, Brazil) connected to a mouthpiece with a 2mm opening to reduce the influence of pressure caused by glottal closure. In a sitting position, each patient performed up to six maneuvers to obtain MIP, from residual volume (RV) to total functional capacity (TFC), considering the best of three maneuvers with < 10% variation between them

SECONDARY OUTCOMES:
Assessment of respiratory mechanics by Optoelectronic Plethysmography | 3 months
  The optoelectronic plethysmography system (OEP) of BTS Bioengineering (Italy) was employed in this study. To that end, a calibration instrument was used, containing three axes connected to reflective markers. This phase does not require participation by the individual to be examined. This creates a three-dimensional model, dividing the thoracoabdominal system into three parts: pulmonary rib cage (RCp), abdominal rib cage (RCa) and the abdomen (AB).
Evaluation of submaximal functional capacity | 3 mounths
  Functional capacity was assessed by the six-minute walk test (6MWT), according to the protocol published by the American Thoracic Society (ATS).
Quality of Life Questionnaire: Minnesota Living With Heart Failure Questionnaire (MLHFQ) | 3 months
  The MLHFQ is a questionnaire validated for the Brazilian population, consisting of 21 questions regarding limitations frequently associated with the extent to which heart failure has affected patient's lives in the previous month. Each question is attributed a value from 0 (zero) to 5 (five), with the highest score indicating worse quality of life. The total score is calculated by adding the 21 items, with a possible interval between 0 and 105.

CONTACTS AND LOCATIONS:
Locations (1):
- Departamento de Fisioterapia-Universidade Federal de pernambuco, Recife, Pernambuco, Brazil

REFERENCES:
- [Result] Chiappa GR, Roseguini BT, Vieira PJ, Alves CN, Tavares A, Winkelmann ER, Ferlin EL, Stein R, Ribeiro JP. Inspiratory muscle training improves blood flow to resting and exercising limbs in patients with chronic heart failure. J Am Coll Cardiol. 2008 Apr 29;51(17):1663-71. doi: 10.1016/j.jacc.2007.12.045. PMID 18436118
- [Result] Olson TP, Beck KC, Johnson BD. Pulmonary function changes associated with cardiomegaly in chronic heart failure. J Card Fail. 2007 Mar;13(2):100-7. doi: 10.1016/j.cardfail.2006.10.018. PMID 17395049